CLINICAL TRIAL: NCT00699699
Title: Assessment of Physical Activity (PF10 Sub Domain of SF-36 Activity Score) and Tolerability in COPD Patients During Treatment With Spiriva® Respimat®
Brief Title: Observational Non-Interventional Study With Spiriva Respimat in COPD Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 205.426
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This observational non-interventional study is designed to demonstrate the improvement of physical function in COPD patients on treatment with Spiriva Respimat and allows adverse events to be recorded and evaluated.

ELIGIBILITY:
Inclusion Criteria:

COPD patients who require treatment with longacting anticholinergic

Exclusion Criteria:

Patients cannot be recruited if any of the general or specific contraindications listed in the Patient information leaflet or the Summary of Product Characteristics applies. Spiriva® Respimat® is contraindicated in patients with hypersensitivity to tiotropium bromide, atropine or its derivatives, e.g. ipratropium or oxitropium or to any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 1280 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (188):
- Germany (188):
  - Boehringer Ingelheim Investigational Site, Aachen
  - Boehringer Ingelheim Investigational Site, Amberg
  - Boehringer Ingelheim Investigational Site, Auerbach
  - Boehringer Ingelheim Investigational Site 1, Augsburg
  - Boehringer Ingelheim Investigational Site 2, Augsburg
  - Boehringer Ingelheim Investigational Site 3, Augsburg
  - Boehringer Ingelheim Investigational Site, Backnang
  - Boehringer Ingelheim Investigational Site, Bad Doberan
  - Boehringer Ingelheim Investigational Site, Bad Kötzing
  - Boehringer Ingelheim Investigational Site, Bad Lippspringe
  - Boehringer Ingelheim Investigational Site, Bad Nauheim
  - Boehringer Ingelheim Investigational Site, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site, Baden-Baden
  - Boehringer Ingelheim Investigational Site 1, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 2, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 1, Berlin
  - Boehringer Ingelheim Investigational Site 2, Berlin
  - Boehringer Ingelheim Investigational Site 3, Berlin
  - Boehringer Ingelheim Investigational Site 4, Berlin
  - Boehringer Ingelheim Investigational Site 5, Berlin
  - Boehringer Ingelheim Investigational Site 6, Berlin
  - Boehringer Ingelheim Investigational Site 7, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site, Bochum
  - Boehringer Ingelheim Investigational Site 1, Bonn
  - Boehringer Ingelheim Investigational Site 2, Bonn
  - Boehringer Ingelheim Investigational Site, Bottrop
  - Boehringer Ingelheim Investigational Site 1, Braunschweig
  - Boehringer Ingelheim Investigational Site 2, Braunschweig
  - Boehringer Ingelheim Investigational Site 3, Braunschweig
  - Boehringer Ingelheim Investigational Site 1, Bremen
  - Boehringer Ingelheim Investigational Site 2, Bremen
  - Boehringer Ingelheim Investigational Site 1, Bremerhaven
  - Boehringer Ingelheim Investigational Site 2, Bremerhaven
  - Boehringer Ingelheim Investigational Site, Burg
  - Boehringer Ingelheim Investigational Site, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site, Celle
  - Boehringer Ingelheim Investigational Site, Cottbus
  - Boehringer Ingelheim Investigational Site, Detmold
  - Boehringer Ingelheim Investigational Site, Dillenburg
  - Boehringer Ingelheim Investigational Site, Donauwörth
  - Boehringer Ingelheim Investigational Site, Dormagen
  - Boehringer Ingelheim Investigational Site, Dorsten
  - Boehringer Ingelheim Investigational Site, Dortmund
  - Boehringer Ingelheim Investigational Site 1, Dresden
  - Boehringer Ingelheim Investigational Site 2, Dresden
  - Boehringer Ingelheim Investigational Site 3, Dresden
  - Boehringer Ingelheim Investigational Site, Duisburg
  - Boehringer Ingelheim Investigational Site, Düren
  - Boehringer Ingelheim Investigational Site 1, Düsseldorf
  - Boehringer Ingelheim Investigational Site 2, Düsseldorf
  - Boehringer Ingelheim Investigational Site 3, Düsseldorf
  - Boehringer Ingelheim Investigational Site 4, Düsseldorf
  - Boehringer Ingelheim Investigational Site 1, Emden
  - Boehringer Ingelheim Investigational Site 2, Emden
  - Boehringer Ingelheim Investigational Site, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site, Erfurt
  - Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site, Euskirchen
  - Boehringer Ingelheim Investigational Site 2, Flensbrug
  - Boehringer Ingelheim Investigational Site 1, Flensburg
  - Boehringer Ingelheim Investigational Site, Frankenthal
  - Boehringer Ingelheim Investigational Site 1, Frankfurt
  - Boehringer Ingelheim Investigational Site 2, Frankfurt
  - Boehringer Ingelheim Investigational Site 3, Frankfurt
  - Boehringer Ingelheim Investigational Site 4, Frankfurt
  - Boehringer Ingelheim Investigational Site, Fürstenfeldbruck
  - Boehringer Ingelheim Investigational Site, Fürstenwalde
  - Boehringer Ingelheim Investigational Site, Fürth
  - Boehringer Ingelheim Investigational Site, Geilenkirchen
  - Boehringer Ingelheim Investigational Site 1, Giessen
  - Boehringer Ingelheim Investigational Site 2, Giessen
  - Boehringer Ingelheim Investigational Site, Grimma
  - Boehringer Ingelheim Investigational Site 1, Gütersloh
  - Boehringer Ingelheim Investigational Site 2, Gütersloh
  - Boehringer Ingelheim Investigational Site, Hainburg
  - Boehringer Ingelheim Investigational Site 1, Hamburg
  - Boehringer Ingelheim Investigational Site 2, Hamburg
  - Boehringer Ingelheim Investigational Site 3, Hamburg
  - Boehringer Ingelheim Investigational Site 4, Hamburg
  - Boehringer Ingelheim Investigational Site 5, Hamburg
  - Boehringer Ingelheim Investigational Site 6, Hamburg
  - Boehringer Ingelheim Investigational Site, Hamm
  - Boehringer Ingelheim Investigational Site 1, Hanover
  - Boehringer Ingelheim Investigational Site 2, Hanover
  - Boehringer Ingelheim Investigational Site 3, Hanover
  - Boehringer Ingelheim Investigational Site 1, Heidelberg
  - Boehringer Ingelheim Investigational Site 2, Heidelberg
  - Boehringer Ingelheim Investigational Site 1, Heilbronn
  - Boehringer Ingelheim Investigational Site 2, Heilbronn
  - Boehringer Ingelheim Investigational Site, Herne
  - Boehringer Ingelheim Investigational Site, Hildburghausen
  - Boehringer Ingelheim Investigational Site, Hilden
  - Boehringer Ingelheim Investigational Site, Hoyerswerda
  - Boehringer Ingelheim Investigational Site, Ibbenbueren
  - Boehringer Ingelheim Investigational Site, Karlsruhe
  - Boehringer Ingelheim Investigational Site 1, Kiel
  - Boehringer Ingelheim Investigational Site 2, Kiel
  - Boehringer Ingelheim Investigational Site 1, Koblenz
  - Boehringer Ingelheim Investigational Site 2, Koblenz
  - Boehringer Ingelheim Investigational Site, Konstanz
  - Boehringer Ingelheim Investigational Site, Königs Wusterhausen
  - Boehringer Ingelheim Investigational Site, Kyritz
  - Boehringer Ingelheim Investigational Site, Leipzig
  - Boehringer Ingelheim Investigational Site 1, Leverkusen
  - Boehringer Ingelheim Investigational Site 2, Leverkusen
  - Boehringer Ingelheim Investigational Site, Limbach-Oberfrohna
  - Boehringer Ingelheim Investigational Site, Lüdenscheid
  - Boehringer Ingelheim Investigational Site, Lüneburg
  - Boehringer Ingelheim Investigational Site 1, Magdeburg
  - Boehringer Ingelheim Investigational Site 2, Magdeburg
  - Boehringer Ingelheim Investigational Site 3, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mannheim
  - Boehringer Ingelheim Investigational Site, Markkleeberg
  - Boehringer Ingelheim Investigational Site, Menden
  - Boehringer Ingelheim Investigational Site, Moers
  - Boehringer Ingelheim Investigational Site, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, Mühlheim
  - Boehringer Ingelheim Investigational Site 1, München
  - Boehringer Ingelheim Investigational Site 2, München
  - Boehringer Ingelheim Investigational Site 3, München
  - Boehringer Ingelheim Investigational Site 4, München
  - Boehringer Ingelheim Investigational Site 5, München
  - Boehringer Ingelheim Investigational Site, Nauen
  - Boehringer Ingelheim Investigational Site, Norderstedt
  - Boehringer Ingelheim Investigational Site, Nordhausen
  - Boehringer Ingelheim Investigational Site, Nordhorn
  - Boehringer Ingelheim Investigational Site 1, Nuremberg
  - Boehringer Ingelheim Investigational Site 2, Nuremberg
  - Boehringer Ingelheim Investigational Site 3, Nuremberg
  - Boehringer Ingelheim Investigational Site 1, Oberhausen
  - Boehringer Ingelheim Investigational Site 2, Oberhausen
  - Boehringer Ingelheim Investigational Site, Oberursel
  - Boehringer Ingelheim Investigational Site 1, Offenbach
  - Boehringer Ingelheim Investigational Site 2, Offenbach
  - Boehringer Ingelheim Investigational Site, Offenburg
  - Boehringer Ingelheim Investigational Site, Olpe
  - Boehringer Ingelheim Investigational Site, Oranienburg
  - Boehringer Ingelheim Investigational Site, Osnabrück
  - Boehringer Ingelheim Investigational Site, Peine
  - Boehringer Ingelheim Investigational Site, Pforzheim
  - Boehringer Ingelheim Investigational Site, Rastatt
  - Boehringer Ingelheim Investigational Site 1, Ratingen
  - Boehringer Ingelheim Investigational Site 2, Ratingen
  - Boehringer Ingelheim Investigational Site, Recklinghausen
  - Boehringer Ingelheim Investigational Site, Remscheid
  - Boehringer Ingelheim Investigational Site, Rostock
  - Boehringer Ingelheim Investigational Site, Roth
  - Boehringer Ingelheim Investigational Site, Rottach-Egern
  - Boehringer Ingelheim Investigational Site, Rudolstadt
  - Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site 1, Saarbrücken
  - Boehringer Ingelheim Investigational Site 2, Saarbrücken
  - Boehringer Ingelheim Investigational Site 3, Saarbrücken
  - Boehringer Ingelheim Investigational Site, Saarlouis
  - Boehringer Ingelheim Investigational Site, Saint Ingbert
  - Boehringer Ingelheim Investigational Site, Salzgitter
  - Boehringer Ingelheim Investigational Site, Schleswig
  - Boehringer Ingelheim Investigational Site, Schmölln
  - Boehringer Ingelheim Investigational Site, Schwandorf in Bayern
  - Boehringer Ingelheim Investigational Site, Sebnitz
  - Boehringer Ingelheim Investigational Site, Siegen
  - Boehringer Ingelheim Investigational Site, Singen
  - Boehringer Ingelheim Investigational Site 1, Solingen
  - Boehringer Ingelheim Investigational Site 2, Solingen
  - Boehringer Ingelheim Investigational Site 3, Solingen
  - Boehringer Ingelheim Investigational Site 4, Solingen
  - Boehringer Ingelheim Investigational Site, Stadthagen
  - Boehringer Ingelheim Investigational Site, Steinhagen
  - Boehringer Ingelheim Investigational Site, Strausberg
  - Boehringer Ingelheim Investigational Site, Stremberg
  - Boehringer Ingelheim Investigational Site, Stuttgart
  - Boehringer Ingelheim Investigational Site, Tauberbischofsheim
  - Boehringer Ingelheim Investigational Site, Tübingen
  - Boehringer Ingelheim Investigational Site 1, Ulm
  - Boehringer Ingelheim Investigational Site 2, Ulm
  - Boehringer Ingelheim Investigational Site 3, Ulm
  - Boehringer Ingelheim Investigational Site, Velbert
  - Boehringer Ingelheim Investigational Site, Waren
  - Boehringer Ingelheim Investigational Site 1, Wiesbaden
  - Boehringer Ingelheim Investigational Site 2, Wiesbaden
  - Boehringer Ingelheim Investigational Site, Wiesloch
  - Boehringer Ingelheim Investigational Site 1, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 2, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site, Witten
  - Boehringer Ingelheim Investigational Site, Wittstock
  - Boehringer Ingelheim Investigational Site, Wolfsburg
  - Boehringer Ingelheim Investigational Site, Zirndorf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time
Started | 1280
Completed | 1223
Not Completed | 57
Not completed — Adverse Event | 36
Not completed — Individual different reasons | 21

BASELINE CHARACTERISTICS:
Arm/Group | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time
Number analyzed (Participants) | 1280
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 500
  Male | 780

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Success as Change From Baseline in Physical Functioning After 6 Weeks
Description: Main efficacy measure was therapeutic success rate defined as an improvement from baseline after 6 weeks by at least 10 score points in the PF-10 (subdomain of SF-36) score (range from 0 to 100, 0 reflects worst and 100 best condition)
Time Frame: Baseline and after 6 weeks of treatment
Population: There were 1230 patients who had evaluable PF-10 measurement at both baseline and after 6 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time
Number analyzed (Participants) | 1230
Percentage of participants | 61.5

2. Secondary Outcome: Change From Baseline in the PF-10 Score After 6 Weeks
Description: Numerical changes in physical functioning (PF-10) after 6 weeks of treatment. PF-10 (subdomain of SF-36) score (range from 0 to 100, 0 reflects worst and 100 best condition)
Time Frame: Baseline and after 6 weeks of treatment
Population: There were 1230 patients who had evaluable PF-10 measurement at both baseline and after 6 weeks
Measure: Mean (Standard Deviation); unit: PF-10 score points
Arm/Group | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time
Number analyzed (Participants) | 1230
PF-10 score points | 13.4 (15.9)

3. Secondary Outcome: Change From Baseline After 6 Weeks in Physician's Global Evaluation (PGE) Form Safety
Description: Changes in Physician's Global Evaluation in physical functioning from baseline after 6 weeks of treatment (measured as 8 point scale with classifications "poor" (1, 2), "satisfactory" (3, 4), "good" (5, 6), and "excellent" (7, 8))
Time Frame: Baseline and after 6 weeks of treatment
Population: There were 1260 patients who had evaluable PGE at both baseline and after 6 weeks
Measure: Mean (Standard Deviation); unit: PGE scale points
Arm/Group | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time
Number analyzed (Participants) | 1260
PGE scale points | 1.1 (1.2)

4. Secondary Outcome: Patients' Satisfaction After 6 Weeks of Treatment
Description: Patients' satisfaction with the Spiriva® Respimat® device after 6 weeks of treatment ("very satisfied", "satisfied", "rather satisfied", "neither satisfied nor "unsatisfied", "rather unsatisfied", "unsatisfied", and "very unsatisfied")
Time Frame: 6 weeks
Population: There were 1260 patients who had evaluable PGE after 6 weeks
Measure: Number; unit: Participants
Arm/Group | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time
Number analyzed (Participants) | 1260
Participants
  Very satisfied | 433
  Satisfied | 551
  Rather satisfied | 145
  Neither / nor | 77
  Rather dissatisfied | 24
  Dissatisfied | 21
  Very dissatisfied | 9

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: There were 1280 patients in the safety population
Arm/Group | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time
Serious Adverse Events (participants affected / at risk) | 6/1280
Other Adverse Events (participants affected / at risk) | 0/1280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva® Respimat® 2 Puffs Once Daily at the Same Time (N=1280)
Tachycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Bronchitis, Infective exacerbation of chronic obstructive airways disease, Urinary tract infection (Infections and infestations) | 3
Bronchial carcinoma, Laryngeal cancer, Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Convulsion (Nervous system disorders) | 1
Azotaemia, Urinary retention (Renal and urinary disorders) | 1
BPH (Reproductive system and breast disorders) | 1
Dyspnoea, Pleural effusion, Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2
Circulatory collapse (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.